CLINICAL TRIAL: NCT00298558
Title: Trial of a Cognitive Intervention for Older Adults
Brief Title: ACTIVE: Advanced Cognitive Training for Independent and Vital Elderly
Acronym: ACTIVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IA0091; U01NR004507 (NIH); U01NR004508 (NIH); U01AG014260 (NIH); U01AG014282 (NIH); U01AG014263 (NIH); U01AG014289 (NIH); U01AG014276 (NIH)
Record Dates: First submitted 2006-02-28; First posted 2006-03-02 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-01

CONDITIONS: Aging; Healthy
Keywords: cognition disorder; cognitive behavior therapy; functional ability
MeSH Terms: conditions — Cognition Disorders | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Memory Training (Active Comparator): Memory training focused on verbal episodic memory. Participants were taught mnemonic strategies for remembering lists and sequences of items, text material, and main ideas and details of stories and other text-based information.
  Interventions: Behavioral: Cognitive Training
- Reasoning Training (Active Comparator): Reasoning training focused on the ability to solve problems that follow a serial pattern. Participants were taught strategies to identify the pattern or sequence required to solve a problem.
  Interventions: Behavioral: Cognitive Training
- Speed of Processing Training (Active Comparator): Speed of processing training focused on visual search and the ability to identify and locate visual information quickly in a divided attention format. Participants practiced increasingly complex speeded tasks on a computer.
  Interventions: Behavioral: Cognitive Training
- Control (Placebo Comparator): This group did not complete any cognitive training interventions
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Cognitive Training — Memory, Reasoning, or Speed of Processing cognitive training interventions

SUMMARY:
The purpose of the ACTIVE study was to test if cognitive training interventions could maintain functional independence in elders by improving basic mental abilities, with follow-up assessments through five years.

DETAILED DESCRIPTION:
ACTIVE was a 4-arm, single-blind, randomized controlled trial. The primary objective of ACTIVE was to test the effectiveness and durability of three distinct cognitive interventions in improving elders' performance on basic measures of cognition and measures of cognitively demanding daily activities (e.g., food preparation, driving, medication use, financial management). These interventions previously had been found successful in improving cognitive abilities under laboratory or small-scale field conditions.

The three interventions shared common design features: 1) equivalent intensity and duration; 2) small group settings in ten 60-75 minute sessions; 3) focus on strategies for solving problems, remembering, or responding quickly to information; 4) modeling and demonstration of strategy usage; 5) practice on exemplar problems; 6) individual and group exercises; 7) feedback on performance; 8) fostering of self-efficacy regarding performance; 9) applying strategies to real-world tasks; 10) individualized training experiences, and 11) social interaction activities. In all three interventions, Sessions 1-5 focused on strategy instruction and exercises to practice the strategy. Sessions 6-10 provided additional practice exercises, but no new strategies were introduced. Content for each of the 10 sessions was scripted in a trainer's manual.

Interventions:

1. Reasoning training focused on inductive reasoning, the ability to solve problems that follow a serial pattern and manifest in executive functioning. Participants were taught strategies to identify the pattern or sequence required to solve a problem. Training exercises involved identifying patterns in both laboratory-type reasoning tasks and in everyday activities, e.g., understanding the pattern in a bus schedule.
2. Memory training focused on verbal episodic memory, which deals with acquisition and retrieval of information acquired in a particular place at a particular time. Participants were taught mnemonic strategies for remembering lists and sequences of items, text material, and main ideas and details of stories and other text-based information. Training exercises involved recalling laboratory-like episodic memory tasks as well as tasks related to everyday activities such as recalling a shopping list.
3. Speed training focused on visual search and the ability to identify and locate visual information quickly in a divided attention format, with and without distractors. Participants practiced speeded tasks on a computer, and were allowed to proceed to more complex tasks, and faster and faster presentation speeds at their own pace.
4. A control group received no training.

In addition, booster training was provided to help participants maintain gains made from initial training and to further improve cognitive skills. Booster training was provided to a random sample of approximately 50% of training participants at 11 and 35-36 months after primary training.

Participant involvement included assessments conducted at baseline, immediately post-intervention, and at 12, 24, 36 and 60 months. Assessments were conducted in individual and group sessions. For participants randomized to intervention groups, the interventions were conducted in small group settings in ten 60-75 minute sessions over a 5-6 week period. These were behavioral interventions with no pharmacologic component. Eleven months after the initial training was provided, booster training was offered, in all three intervention arms, to a randomly selected 60% of initially trained subjects. Booster training was delivered in four 75-minute sessions over a 2-3 week period.

The primary study hypotheses were:

* Each training group will perform better than the other training and control groups on their respective primary and proximal outcomes
* Those groups that received booster training will perform better than those that did not receive booster training on their respective primary and proximal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* Mini-Mental State Examination (MMSE) score 23 or greater
* Vision scored greater than 20/50
* Minimal dependence in hygiene, bathing, and dressing

Exclusion Criteria:

* Significant decline in cognitive skills, physical abilities, or functional independence
* Inability to complete study activities as evidenced by MMSE and vision scores lower than Inclusion Criteria requirement
* Diagnosis of Alzheimer's disease
* Stroke in previous 12 months
* Cancer with limited life expectance
* Current chemotherapy or radiation treatment
* Communication problems
* Planned move from study area
* Scheduling conflicts that would preclude participation in study activities
* Prior involvement in similar cognitive training studies

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2832 (Actual)
Dates: Start 1998-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karlene Ball, PhD, Principal Investigator — University of Alabama at Birmingham; Frederick Unverzagt, PhD, Principal Investigator — Indiana University; George Rebok, PhD, Principal Investigator — Johns Hopkins University; John Morris, PhD, Principal Investigator — Hebrew Senior Life; Sharon L. Tennstedt, PhD, Principal Investigator — Carelon Research; Michael Marsiske, PhD, Principal Investigator — Wayne State University; Sherry Willis, PhD, Principal Investigator — Penn State University
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Johns Hopkins University, Cumberland, Maryland
  - Hebrew Rehabilitation Center for the Aged, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Pennsylvania State University, University Park, Pennsylvania

REFERENCES:
- [Background] Jobe JB, Smith DM, Ball K, Tennstedt SL, Marsiske M, Willis SL, Rebok GW, Morris JN, Helmers KF, Leveck MD, Kleinman K. ACTIVE: a cognitive intervention trial to promote independence in older adults. Control Clin Trials. 2001 Aug;22(4):453-79. doi: 10.1016/s0197-2456(01)00139-8. PMID 11514044
- [Background] Jones RN, Rosenberg AL, Morris JN, Allaire JC, McCoy KJ, Marsiske M, Kleinman KP, Rebok GW, Malloy PF. A growth curve model of learning acquisition among cognitively normal older adults. Exp Aging Res. 2005 Jul-Sep;31(3):291-312. doi: 10.1080/03610730590948195. PMID 16036723
- [Background] Kuo HK, Jones RN, Milberg WP, Tennstedt S, Talbot L, Morris JN, Lipsitz LA. Cognitive function in normal-weight, overweight, and obese older adults: an analysis of the Advanced Cognitive Training for Independent and Vital Elderly cohort. J Am Geriatr Soc. 2006 Jan;54(1):97-103. doi: 10.1111/j.1532-5415.2005.00522.x. PMID 16420204
- [Background] Diehl M, Marsiske M, Horgas AL, Rosenberg A, Saczynski JS, Willis SL. The Revised Observed Tasks of Daily Living: A Performance-Based Assessment of Everyday Problem Solving in Older Adults. J Appl Gerontol. 2005;24(3):211-230. doi: 10.1177/0733464804273772. PMID 18160968
- [Background] Wadley VG, Crowe M, Marsiske M, Cook SE, Unverzagt FW, Rosenberg AL, Rexroth D. Changes in everyday function in individuals with psychometrically defined mild cognitive impairment in the Advanced Cognitive Training for Independent and Vital Elderly Study. J Am Geriatr Soc. 2007 Aug;55(8):1192-8. doi: 10.1111/j.1532-5415.2007.01245.x. PMID 17661957
- [Background] Cook SE, Marsiske M, Thomas KR, Unverzagt FW, Wadley VG, Langbaum JB, Crowe M. Identification of mild cognitive impairment in ACTIVE: algorithmic classification and stability. J Int Neuropsychol Soc. 2013 Jan;19(1):73-87. doi: 10.1017/S1355617712000938. Epub 2012 Oct 25. PMID 23095218
- [Background] Owsley C, Sloane M, McGwin G Jr, Ball K. Timed instrumental activities of daily living tasks: relationship to cognitive function and everyday performance assessments in older adults. Gerontology. 2002 Jul-Aug;48(4):254-65. doi: 10.1159/000058360. PMID 12053117
- [Background] Gallo JJ, Rebok GW, Tennsted S, Wadley VG, Horgas A; Advanced Cognitive Training for Independent and Vital Elderly (Active) Study Investigators. Linking depressive symptoms and functional disability in late life. Aging Ment Health. 2003 Nov;7(6):469-80. doi: 10.1080/13607860310001594736. PMID 14578009
- [Background] Caskie GI, Willis SL. Congruence of self-reported medications with pharmacy prescription records in low-income older adults. Gerontologist. 2004 Apr;44(2):176-85. doi: 10.1093/geront/44.2.176. PMID 15075414
- [Background] Edwards JD, Ross LA, Wadley VG, Clay OJ, Crowe M, Roenker DL, Ball KK. The useful field of view test: normative data for older adults. Arch Clin Neuropsychol. 2006 May;21(4):275-86. doi: 10.1016/j.acn.2006.03.001. Epub 2006 May 15. PMID 16704918
- [Background] Wolinsky FD, Unverzagt FW, Smith DM, Jones R, Wright E, Tennstedt SL. The effects of the ACTIVE cognitive training trial on clinically relevant declines in health-related quality of life. J Gerontol B Psychol Sci Soc Sci. 2006 Sep;61(5):S281-7. doi: 10.1093/geronb/61.5.s281. PMID 16960242
- [Background] Crowe M, Andel R, Wadley V, Cook S, Unverzagt F, Marsiske M, Ball K. Subjective cognitive function and decline among older adults with psychometrically defined amnestic MCI. Int J Geriatr Psychiatry. 2006 Dec;21(12):1187-92. doi: 10.1002/gps.1639. PMID 16955448
- [Background] Kuo HK, Jones RN, Milberg WP, Tennstedt S, Talbot L, Morris JN, Lipsitz LA. Effect of blood pressure and diabetes mellitus on cognitive and physical functions in older adults: a longitudinal analysis of the advanced cognitive training for independent and vital elderly cohort. J Am Geriatr Soc. 2005 Jul;53(7):1154-61. doi: 10.1111/j.1532-5415.2005.53368.x. PMID 16108933
- [Background] Wolinsky FD, Unverzagt FW, Smith DM, Jones R, Stoddard A, Tennstedt SL. The ACTIVE cognitive training trial and health-related quality of life: protection that lasts for 5 years. J Gerontol A Biol Sci Med Sci. 2006 Dec;61(12):1324-9. doi: 10.1093/gerona/61.12.1324. PMID 17234829
- [Background] Ball K, Edwards JD, Ross LA. The impact of speed of processing training on cognitive and everyday functions. J Gerontol B Psychol Sci Soc Sci. 2007 Jun;62 Spec No 1:19-31. doi: 10.1093/geronb/62.special_issue_1.19. PMID 17565162
- [Background] Rebok GW, Carlson MC, Langbaum JB. Training and maintaining memory abilities in healthy older adults: traditional and novel approaches. J Gerontol B Psychol Sci Soc Sci. 2007 Jun;62 Spec No 1:53-61. doi: 10.1093/geronb/62.special_issue_1.53. PMID 17565165
- [Background] Unverzagt FW, Kasten L, Johnson KE, Rebok GW, Marsiske M, Koepke KM, Elias JW, Morris JN, Willis SL, Ball K, Rexroth DF, Smith DM, Wolinsky FD, Tennstedt SL. Effect of memory impairment on training outcomes in ACTIVE. J Int Neuropsychol Soc. 2007 Nov;13(6):953-60. doi: 10.1017/S1355617707071512. PMID 17942013
- [Background] Edwards JD, Ross LA, Ackerman ML, Small BJ, Ball KK, Bradley S, Dodson JE. Longitudinal predictors of driving cessation among older adults from the ACTIVE clinical trial. J Gerontol B Psychol Sci Soc Sci. 2008 Jan;63(1):P6-12. doi: 10.1093/geronb/63.1.p6. PMID 18332196
- [Background] Morgan AA, Marsiske M, Whitfield KE. Characterizing and explaining differences in cognitive test performance between african american and European American older adults. Exp Aging Res. 2008 Jan-Mar;34(1):80-100. doi: 10.1080/03610730701776427. PMID 18189169
- [Background] Vance DE, Ross LA, Crowe MG, Wadley VG, Edwards JD, Ball KK. THE RELATIONSHIP OF MEMORY, REASONING, AND SPEED OF PROCESSING ON FALLING AMONG OLDER ADULTS. Phys Occup Ther Geriatr. 2008;27(3):212-228. doi: 10.1080/02703180802377123. PMID 20216922
- [Background] Ackerman ML, Edwards JD, Ross LA, Ball KK, Lunsman M. Examination of cognitive and instrumental functional performance as indicators for driving cessation risk across 3 years. Gerontologist. 2008 Dec;48(6):802-10. doi: 10.1093/geront/48.6.802. PMID 19139253
- [Background] Langbaum JB, Rebok GW, Bandeen-Roche K, Carlson MC. Predicting memory training response patterns: results from ACTIVE. J Gerontol B Psychol Sci Soc Sci. 2009 Jan;64(1):14-23. doi: 10.1093/geronb/gbn026. Epub 2009 Feb 4. PMID 19196693
- [Background] Tucker-Drob EM, Johnson KE, Jones RN. The cognitive reserve hypothesis: a longitudinal examination of age-associated declines in reasoning and processing speed. Dev Psychol. 2009 Mar;45(2):431-46. doi: 10.1037/a0014012. PMID 19271829
- [Background] Ross LA, Clay OJ, Edwards JD, Ball KK, Wadley VG, Vance DE, Cissell GM, Roenker DL, Joyce JJ. Do older drivers at-risk for crashes modify their driving over time? J Gerontol B Psychol Sci Soc Sci. 2009 Mar;64(2):163-70. doi: 10.1093/geronb/gbn034. Epub 2009 Feb 4. PMID 19196692
- [Background] Wolinsky FD, Vander Weg MW, Martin R, Unverzagt FW, Ball KK, Jones RN, Tennstedt SL. The effect of speed-of-processing training on depressive symptoms in ACTIVE. J Gerontol A Biol Sci Med Sci. 2009 Apr;64(4):468-72. doi: 10.1093/gerona/gln044. Epub 2009 Jan 30. PMID 19181719
- [Background] Wolinsky FD, Mahncke HW, Kosinski M, Unverzagt FW, Smith DM, Jones RN, Stoddard A, Tennstedt SL. The ACTIVE cognitive training trial and predicted medical expenditures. BMC Health Serv Res. 2009 Jun 29;9:109. doi: 10.1186/1472-6963-9-109. PMID 19558724
- [Background] Unverzagt FW, Smith DM, Rebok GW, Marsiske M, Morris JN, Jones R, Willis SL, Ball K, King JW, Koepke KM, Stoddard A, Tennstedt SL. The Indiana Alzheimer Disease Center's Symposium on Mild Cognitive Impairment. Cognitive training in older adults: lessons from the ACTIVE Study. Curr Alzheimer Res. 2009 Aug;6(4):375-83. doi: 10.2174/156720509788929345. PMID 19689237
- [Background] Wolinsky FD, Mahncke HW, Weg MW, Martin R, Unverzagt FW, Ball KK, Jones RN, Tennstedt SL. The ACTIVE cognitive training interventions and the onset of and recovery from suspected clinical depression. J Gerontol B Psychol Sci Soc Sci. 2009 Sep;64(5):577-85. doi: 10.1093/geronb/gbp061. Epub 2009 Jul 17. PMID 19617456
- [Background] Edwards JD, Lunsman M, Perkins M, Rebok GW, Roth DL. Driving cessation and health trajectories in older adults. J Gerontol A Biol Sci Med Sci. 2009 Dec;64(12):1290-5. doi: 10.1093/gerona/glp114. Epub 2009 Aug 12. PMID 19675177
- [Background] Edwards JD, Delahunt PB, Mahncke HW. Cognitive speed of processing training delays driving cessation. J Gerontol A Biol Sci Med Sci. 2009 Dec;64(12):1262-7. doi: 10.1093/gerona/glp131. Epub 2009 Sep 2. PMID 19726665
- [Background] Kvale EA, Clay OJ, Ross-Meadows LA, McGee JS, Edwards JD, Unverzagt FW, Ritchie CS, Ball KK. Cognitive speed of processing and functional declines in older cancer survivors: an analysis of data from the ACTIVE trial. Eur J Cancer Care (Engl). 2010 Jan 1;19(1):110-7. doi: 10.1111/j.1365-2354.2008.01018.x. Epub 2009 Aug 26. PMID 19709169
- [Background] Wolinsky FD, Mahncke H, Vander Weg MW, Martin R, Unverzagt FW, Ball KK, Jones RN, Tennstedt SL. Speed of processing training protects self-rated health in older adults: enduring effects observed in the multi-site ACTIVE randomized controlled trial. Int Psychogeriatr. 2010 May;22(3):470-8. doi: 10.1017/S1041610209991281. Epub 2009 Dec 15. PMID 20003628
- [Background] O'Connor ML, Edwards JD, Wadley VG, Crowe M. Changes in mobility among older adults with psychometrically defined mild cognitive impairment. J Gerontol B Psychol Sci Soc Sci. 2010 May;65B(3):306-16. doi: 10.1093/geronb/gbq003. Epub 2010 Feb 10. PMID 20147739
- [Background] Yen YC, Rebok GW, Gallo JJ, Jones RN, Tennstedt SL. Depressive symptoms impair everyday problem-solving ability through cognitive abilities in late life. Am J Geriatr Psychiatry. 2011 Feb;19(2):142-50. doi: 10.1097/JGP.0b013e3181e89894. PMID 20808123
- [Background] Wolinsky FD, Vander Weg MW, Martin R, Unverzagt FW, Willis SL, Marsiske M, Rebok GW, Morris JN, Ball KK, Tennstedt SL. Does cognitive training improve internal locus of control among older adults? J Gerontol B Psychol Sci Soc Sci. 2010 Sep;65(5):591-8. doi: 10.1093/geronb/gbp117. Epub 2009 Dec 11. PMID 20008028
- [Background] Aiken Morgan AT, Marsiske M, Dzierzewski JM, Jones RN, Whitfield KE, Johnson KE, Cresci MK. Race-related cognitive test bias in the active study: a mimic model approach. Exp Aging Res. 2010 Oct;36(4):426-52. doi: 10.1080/0361073X.2010.507427. PMID 20845121
- [Background] Gross AL, Rebok GW, Unverzagt FW, Willis SL, Brandt J. Word list memory predicts everyday function and problem-solving in the elderly: results from the ACTIVE cognitive intervention trial. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2011 Mar;18(2):129-46. doi: 10.1080/13825585.2010.516814. Epub 2010 Nov 10. PMID 21069610
- [Background] Ball K, Edwards JD, Ross LA, McGwin G Jr. Cognitive training decreases motor vehicle collision involvement of older drivers. J Am Geriatr Soc. 2010 Nov;58(11):2107-13. doi: 10.1111/j.1532-5415.2010.03138.x. PMID 21054291
- [Background] Parisi JM, Gross AL, Rebok GW, Saczynski JS, Crowe M, Cook SE, Langbaum JB, Sartori A, Unverzagt FW. Modeling change in memory performance and memory perceptions: findings from the ACTIVE study. Psychol Aging. 2011 Sep;26(3):518-24. doi: 10.1037/a0022458. PMID 21463064
- [Background] O'Connor ML, Edwards JD, Small BJ, Andel R. Patterns of level and change in self-reported driving behaviors among older adults: who self-regulates? J Gerontol B Psychol Sci Soc Sci. 2012 Jul;67(4):437-46. doi: 10.1093/geronb/gbr122. Epub 2011 Dec 1. PMID 22138270
- [Background] Gross AL, Rebok GW. Memory training and strategy use in older adults: results from the ACTIVE study. Psychol Aging. 2011 Sep;26(3):503-17. doi: 10.1037/a0022687. PMID 21443356
- [Background] Gross AL, Rebok GW, Unverzagt FW, Willis SL, Brandt J. Cognitive predictors of everyday functioning in older adults: results from the ACTIVE Cognitive Intervention Trial. J Gerontol B Psychol Sci Soc Sci. 2011 Sep;66(5):557-66. doi: 10.1093/geronb/gbr033. Epub 2011 May 9. PMID 21558167
- [Background] Unverzagt FW, Guey LT, Jones RN, Marsiske M, King JW, Wadley VG, Crowe M, Rebok GW, Tennstedt SL. ACTIVE cognitive training and rates of incident dementia. J Int Neuropsychol Soc. 2012 Jul;18(4):669-77. doi: 10.1017/S1355617711001470. Epub 2012 Mar 9. PMID 22400989
- [Background] Sisco SM, Marsiske M. Neighborhood Influences on Late Life Cognition in the ACTIVE Study. J Aging Res. 2012;2012:435826. doi: 10.1155/2012/435826. Epub 2012 Aug 26. PMID 22966458
- [Background] Gross AL, Inouye SK, Rebok GW, Brandt J, Crane PK, Parisi JM, Tommet D, Bandeen-Roche K, Carlson MC, Jones RN. Parallel but not equivalent: challenges and solutions for repeated assessment of cognition over time. J Clin Exp Neuropsychol. 2012;34(7):758-72. doi: 10.1080/13803395.2012.681628. Epub 2012 Apr 30. PMID 22540849
- [Background] Gross AL, Rebok GW, Brandt J, Tommet D, Marsiske M, Jones RN. Modeling learning and memory using verbal learning tests: results from ACTIVE. J Gerontol B Psychol Sci Soc Sci. 2013 Mar;68(2):153-67. doi: 10.1093/geronb/gbs053. Epub 2012 Aug 28. PMID 22929389
- [Background] Sartori AC, Wadley VG, Clay OJ, Parisi JM, Rebok GW, Crowe M. The relationship between cognitive function and life space: the potential role of personal control beliefs. Psychol Aging. 2012 Jun;27(2):364-74. doi: 10.1037/a0025212. Epub 2011 Aug 29. PMID 21875217
- [Background] Lin F, Chen DG, Vance DE, Ball KK, Mapstone M. Longitudinal relationships between subjective fatigue, cognitive function, and everyday functioning in old age. Int Psychogeriatr. 2013 Feb;25(2):275-85. doi: 10.1017/S1041610212001718. Epub 2012 Oct 19. PMID 23083533
- [Result] Ball K, Berch DB, Helmers KF, Jobe JB, Leveck MD, Marsiske M, Morris JN, Rebok GW, Smith DM, Tennstedt SL, Unverzagt FW, Willis SL; Advanced Cognitive Training for Independent and Vital Elderly Study Group. Effects of cognitive training interventions with older adults: a randomized controlled trial. JAMA. 2002 Nov 13;288(18):2271-81. doi: 10.1001/jama.288.18.2271. PMID 12425704
- [Result] Willis SL, Tennstedt SL, Marsiske M, Ball K, Elias J, Koepke KM, Morris JN, Rebok GW, Unverzagt FW, Stoddard AM, Wright E; ACTIVE Study Group. Long-term effects of cognitive training on everyday functional outcomes in older adults. JAMA. 2006 Dec 20;296(23):2805-14. doi: 10.1001/jama.296.23.2805. PMID 17179457
- [Derived] Phillips CB, McVey A, Sprague BN, Cooper K, Stephan AT, Ross LA. Predictive Utility of Four Instrumental Activities of Daily Living Assessments and Cognitive Status Changes Among Cognitively In-Tact Older Adults. J Aging Health. 2025 Dec;37(10):683-693. doi: 10.1177/08982643241297193. Epub 2024 Nov 9. PMID 39520262
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] Sprague BN, Ross LA, Ball KK. Does Cognitive Training Reduce Falls across Ten Years?: Data from the ACTIVE Trial. Int J Environ Res Public Health. 2023 Mar 11;20(6):4941. doi: 10.3390/ijerph20064941. PMID 36981850
- [Derived] Bell TR, Sprague BN, Ross LA. Longitudinal associations of pain and cognitive decline in community-dwelling older adults. Psychol Aging. 2022 Sep;37(6):715-730. doi: 10.1037/pag0000699. Epub 2022 Jul 28. PMID 35901382
- [Derived] Chamberlain JD, Sprague BN, Ross LA. Age- and Time-Varying Associations Between Subjective Health and Episodic Memory in Older Adults. J Gerontol B Psychol Sci Soc Sci. 2022 Apr 1;77(4):673-682. doi: 10.1093/geronb/gbab142. PMID 34329436
- [Derived] Clark DO, Xu H, Callahan CM, Unverzagt FW. Does Body Mass Index Modify Memory, Reasoning, and Speed of Processing Training Effects in Older Adults. Obesity (Silver Spring). 2016 Nov;24(11):2319-2326. doi: 10.1002/oby.21631. PMID 27804270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from March 1998 through October 1999 at six metropolitan field centers: University of Alabama at Birmingham, Boston Hebrew Rehabilitation Center for Aged (now Hebrew Senior Life), Indiana University School of Medicine, Johns Hopkins University, Pennsylvania State University, and Wayne State University.
Pre-assignment Details: Eligibility and demographics were gathered at telephone screening.Health history, physical status, functional status, mental status, cognitive and function measures were gathered via in-person exams in individual and small-group formats at baseline.Eligible subjects were randomly assigned to one of three interventions or no-contact control group.
Period: Baseline
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Started | 711 | 705 | 712 | 704
Completed | 711 | 705 | 712 | 704
Not Completed | 0 | 0 | 0 | 0
Period: Intervention
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Started | 711 | 705 | 712 | 704
Completed | 620 | 627 | 637 | 285
Not Completed | 91 | 78 | 75 | 419
Period: Immediate Post Test
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Started | 711 | 705 | 712 | 704
Completed | 640 | 629 | 653 | 639
Not Completed | 71 | 76 | 59 | 65
Period: Booster
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Started | 372 | 371 | 370 | 0
Completed | 283 | 301 | 295 | 0
Not Completed | 89 | 70 | 75 | 0
Period: 1st Annual (A1)
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Started | 640 | 629 | 653 | 639
Completed | 585 | 566 | 601 | 584
Not Completed | 55 | 63 | 52 | 55
Period: 2nd Annual (A2)
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Started | 585 | 566 | 601 | 584
Completed | 563 | 555 | 574 | 552
Not Completed | 22 | 11 | 27 | 32
Period: 3rd Annual Booster
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Started | 372 | 371 | 370 | 0
Completed | 250 | 243 | 230 | 0
Not Completed | 122 | 128 | 140 | 0
Period: 3rd Annual (A3) and 5th Annual (A5)
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Started | 563 | 555 | 574 | 552
Completed | 472 | 469 | 490 | 448
Not Completed | 91 | 86 | 84 | 104
Period: 10th Annual (A10)
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Started | 472 | 469 | 490 | 448
Completed | 300 | 316 | 319 | 285
Not Completed | 172 | 153 | 171 | 163

BASELINE CHARACTERISTICS:
Population: Of 2832 randomized subjects, 30 subjects were randomized inappropriately in violation of the protocol and excluded from the analysis. Therefore, 2802 subjects were used for the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control | Total
Number analyzed (Participants) | 703 | 699 | 702 | 698 | 2802
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 703 | 699 | 702 | 698 | 2802
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (6.02) | 73.5 (5.76) | 73.4 (5.78) | 74.0 (6.05) | 73.6 (5.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 537 | 537 | 538 | 514 | 2126
  Male | 166 | 162 | 164 | 184 | 676
Region of Enrollment [Number; unit: participants]
  United States | 703 | 699 | 702 | 698 | 2802

OUTCOME MEASURES:

1. Primary Outcome: Changes in Cognitive Abilities of Memory From Baseline to Year 10
Description: Memory outcome was computed as the summation of Rey Auditory-Verbal Learning Test (AVLT), the Hopkins Verbal Learning Test (HVLT), and the Rivermead Behavioral Paragraph Recall test immediate recall. The possible range of the memory outcome is 0 to 132. Higher values represent a better outcome. Changes in outcome were computed as "10 year minus baseline" and the negative values indicate the decline from baseline.
Time Frame: Up to 10 years
Population: Of the randomized subjects, 943 subjects who had the memory outcome at year 10 were used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Number analyzed (Participants) | 231 | 248 | 248 | 216
units on a scale | -10.6 (28.3) | -11.2 (26.3) | -12.7 (25.5) | -9.4 (29.6)
Statistical Analysis 1: Comparison: Memory Training vs Control; Effect size was defined as training improvement from baseline to year 10 minus control improvement from baseline to year 10 divided by the intrasubject standard deviation (SD) of the composite score. Positive effect sizes indicate improvement; Test type: Superiority or Other; p = 0.43, Mixed Models Analysis; The blom transformation was used to reduce skewness in the measures. The design factors and baseline covariates were controlled in the model; Effect Size = 0.06, 99% CI 2-sided [-0.14 to 0.27] — Blom transformed outcome was used and the design factors and baseline covariates were controlled in the model to get the adjusted means. After that, the effect size (defined in the Additional details) was calculated using the adjusted means and SD
Statistical Analysis 2: Comparison: Reasoning Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.17, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = -0.11, 99% CI 2-sided [-0.31 to 0.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Speed of Processing Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.52, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = -0.05, 99% CI 2-sided [-0.25 to 0.15] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Changes in Health-related Quality of Life (HRQol), Driving Function, Health Service Use
Description: To determine if the cognitive interventions have beneficial effects on the distal outcomes of driving safety, personal care activities of daily living, health service utilization, and mortality.
Time Frame: 10th Year
Reporting Status: Not Posted

3. Secondary Outcome: Examine Health, Genetic and Cognitive Moderators
Description: To examine heath, genetic, and cognitive moderators (including cardiovascular disease,diabetes, depression, Apolipoprotein E (APOE) genotype, and low cognition and engagement) in individual response to training.
Time Frame: 10th Year
Reporting Status: Not Posted

4. Primary Outcome: Changes in Cognitive Abilities of Reasoning From Baseline to Year 10
Description: Reasoning outcome was computed as the summation of total correct for Letter Series, Letter Sets, and Word Series. The possible range of the reasoning outcome is 0 to 75. Higher values represent a better outcome. Changes in outcome were computed as "10 year minus baseline" and the negative values indicate the decline from baseline.
Time Frame: Up to 10 years
Population: Of the randomized subjects, 938 subjects who had the reasoning outcome at year 10 were used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Number analyzed (Participants) | 230 | 246 | 248 | 214
units on a scale | -3.23 (8.61) | -0.049 (7.91) | -3.94 (8.34) | -3.04 (8.02)
Statistical Analysis 1: Comparison: Memory Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.69, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = -0.02, 99% CI 2-sided [-0.17 to 0.12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Reasoning Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = 0.23, 99% CI 2-sided [0.09 to 0.38] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Speed of Processing Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.27, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = -0.06, 99% CI 2-sided [-0.20 to 0.08] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Estimate the Effects of ACTIVE Training to General Population
Description: To estimate and project the effects of ACTIVE training to the general population of older adults by linking the measures and outcomes of ACTIVE to the Health and Retirement Study(and its subsidiary studies), a population-based, nationally-representative cohort.
Time Frame: 10th Year
Reporting Status: Not Posted

6. Primary Outcome: Changes in Cognitive Abilities of Speed of Processing From Baseline to Year 10
Description: Speed of processing outcome was computed as the summation of three Useful Field of View tasks requiring identification and localization of information, with 75% accuracy, under varying levels of cognitive demand. For the analysis, the reversed score was used and the possible range of the reversed speed of processing outcome is 0 to 1500. Higher values for the reversed scores represent a better outcome. Changes in outcome were computed as "10 year minus baseline" and the negative values indicate the decline from baseline.
Time Frame: Up to 10 years
Population: Of the randomized subjects, 879 subjects who had the speed outcome at year 10 were used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Number analyzed (Participants) | 216 | 231 | 229 | 203
units on a scale | -144.4 (228.6) | -126.2 (253.6) | 24.3 (252.1) | -123.3 (277.7)
Statistical Analysis 1: Comparison: Memory Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.45, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = -0.07, 99% CI 2-sided [-0.29 to 0.16] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Reasoning Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.95, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = 0.005, 99% CI 2-sided [-0.22 to 0.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Speed of Processing Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = 0.66, 99% CI 2-sided [0.43 to 0.88] — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: Changes in Instrumental Activities of Daily Living (IADL) Difficulty From Baseline to Year 10
Description: The self-reported measure of everyday IADL function was the summation of the IADL difficulty sub-scores from the Minimum Dataset - Home Care (MDS-HC) which assesses performance in the past 7 days on 19 daily tasks spanning meal preparation, housework, finances, health care, telephone, shopping, travel, and need for assistance in dressing, personal hygiene, and bathing. For the analysis, the reversed score was used and the possible range of the reversed everyday IADL function outcome is 0 to 38. Higher values for the reversed scores represent a better outcome. Changes in outcome were computed as "10 year minus baseline" and the negative values indicate the decline from baseline.
Time Frame: Up to 10 years
Population: Of the randomized subjects, 1211 subjects who had the IADL outcome at year 10 were used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Number analyzed (Participants) | 297 | 314 | 316 | 284
units on a scale | -3.05 (7.38) | -2.66 (6.31) | -2.34 (5.62) | -3.61 (7.67)
Statistical Analysis 1: Comparison: Memory Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = 0.48, 99% CI 2-sided [0.12 to 0.84] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Reasoning Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = 0.38, 99% CI 2-sided [0.02 to 0.74] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Speed of Processing Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = 0.36, 99% CI 2-sided [0.01 to 0.72] — [estimate comment as in outcome 1, analysis 1]

8. Primary Outcome: Changes in Everyday Problem Solving From Baseline to Year 10
Description: Everyday Problem Solving was computed as the summation of the Everyday Problems Test (EPT) and Observed Tasks of Daily Living (OTDL). The possible range of the everyday problem solving outcome is 0 to 56. Higher values represent a better outcome. Changes in outcome were computed as "10 year minus baseline" and the negative values indicate the decline from baseline.
Time Frame: Up to 10 years
Population: Of the randomized subjects, 1104 subjects who had the everyday problem solving outcome at year 10 were used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Number analyzed (Participants) | 270 | 290 | 295 | 249
units on a scale | -6.10 (9.75) | -5.58 (9.56) | -5.98 (9.32) | -5.67 (9.85)
Statistical Analysis 1: Comparison: Memory Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.97, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = 0.004, 99% CI 2-sided [-0.23 to 0.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Reasoning Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.86, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = -0.02, 99% CI 2-sided [-0.25 to 0.22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Speed of Processing Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.93, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = 0.008, 99% CI 2-sided [-0.23 to 0.24] — [estimate comment as in outcome 1, analysis 1]

9. Primary Outcome: Changes in Everyday Speed of Processing From Baseline to Year 10
Description: Everyday Speed of processing was computed as the summation of Complex Reaction Time (CRT) and Timed IADL (TIADL). For the analysis, the reversed score was used and the possible range of the reversed everyday speed of processing outcome is -3 to 100. Higher values for the reversed scores represent a better outcome. Changes in outcome were computed as "10 year minus baseline" and the negative values indicate the decline from baseline.
Time Frame: Up to 10 years
Population: Of the randomized subjects, 938 subjects who had the everyday speed of processing outcome at year 10 were used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Number analyzed (Participants) | 229 | 249 | 245 | 215
units on a scale | -1.53 (2.17) | -1.39 (1.88) | -1.47 (1.98) | -1.42 (1.78)
Statistical Analysis 1: Comparison: Memory Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.78, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = 0.02, 99% CI 2-sided [-0.19 to 0.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Reasoning Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.96, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = -0.004, 99% CI 2-sided [-0.21 to 0.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Speed of Processing Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.56, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Effect Size = -0.05, 99% CI 2-sided [-0.26 to 0.16] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Memory Training | Reasoning Training | Speed of Processing Training | Control
Serious Adverse Events (participants affected / at risk) | 0/711 | 0/705 | 0/712 | 0/704
Other Adverse Events (participants affected / at risk) | 0/711 | 0/705 | 0/712 | 0/704

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.